CLINICAL TRIAL: NCT03681366
Title: Myopia Control Using Optimized Optical Defocus in Schoolchildren - a Randomized Double Masked Control Trial
Brief Title: Myopia Control Using Optimized Optical Defocus RCTs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Principal Investigator, Carly Lam, Professor, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HSEARS20180711001
Record Dates: First submitted 2018-09-20; First posted 2018-09-24 (Actual); Last update posted 2022-08-24 (Actual); Status verified 2022-08

CONDITIONS: Myopia
Keywords: myopia; Myopic Defocus; contact lens; myopia control
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Double masked design:
  The investigator(s) who were responsible for refracting and performing relevant ocular data measurement were masked from the grouping of the subjects.
  The unmasked investigator(s) were responsible for group allocation, spectacle-dispensing work, measuring lens visual performance, record keeping, data entry and compliance checking. Data input was carefully checked by the unmasked investigator and the other researchers independently.
  The children and their parents were also masked to group allocation until the data analysis was completed.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Single vision soft contact lens (No Intervention): single vision, spherical soft contact lens
- DISC3.5 Plus lens (Experimental): A soft contact lens that comprises of simultaneous distance optical prescription and myopic defocus areas.
  Interventions: Device: DISC3.5 plus

INTERVENTIONS:
Device: DISC3.5 plus — The Defocus Incorporated Soft 3.5 Plus Contact Lens (DISC3.5 Plus) is a soft contact lens that comprises of simultaneous distance optical prescription and myopic defocus areas.
  Arms: DISC3.5 Plus lens

SUMMARY:
The aims of the study is to evaluate whether the DISC3.5 Plus contact lens will slow myopia progression and axial length growth in myopic children as compared with single vision soft contact lenses.

DETAILED DESCRIPTION:
The purpose of the current study is to evaluate whether the DISC3.5 Plus contact lens will slow myopia progression and axial length growth in myopic children as compared with single vision soft contact lenses.

The Defocus Incorporated Soft 3.5 Plus Contact Lens (DISC3.5 Plus) is a soft contact lens that comprises of simultaneous distance optical prescription and myopic defocus areas.

The efficacy of the DISC3.5 Plus lens in slowing myopia progression (change in refractive error) will be compared to a spherical (front and back surface) single vision soft contact lenses in this one-year prospective, randomised and double-masked clinical trial. The hypothesis of this study is that the DISC3.5 Plus will slow myopia progression more than spherical single vision soft contact lenses.

ELIGIBILITY:
Inclusion Criteria:

* Age at enrolment: 8-13 year; Hong Kong Chinese
* Spherical equivalent refractions (SER): -1.00 to -5.00D
* Astigmatism: -1.00D or less
* Anisometropia: 1.25D or less
* Spectacle corrected monocular visual acuity (VA): 0.0 logMAR or better
* Contact lens corrected monocular VA: 0.1 logMAR or better
* Normal binocular function
* Willingness to wear contact lenses regularly
* Parents' understanding and acceptance of random allocation of grouping and masking

Exclusion Criteria:

* Prior myopia control treatment, e.g. orthokeratology, defocus soft contact lenses, progressive addition lenses, bifocal lenses, drugs (e.g. atropine), etc.
* Strabismus or decompensated phoria (checked by cover test at far and near in screening)
* Known contraindications for contact lens wear
* Have any ocular and systemic diseases and abnormalities that might affect visual function or refractive development

Ages: 8 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 167 (Actual)
Dates: Start 2018-10-25 (Actual); Primary Completion 2021-05-08 (Actual); Study Completion 2022-06-24 (Actual)

PRIMARY OUTCOMES:
Cycloplegic Refraction Change in SER | 12 months
  Change in cycloplegic autorefraction in spherical equivalent (SER)

SECONDARY OUTCOMES:
Axial length | 12 months
  Axial length (mm) was measured after cycloplegia

CONTACTS AND LOCATIONS:
Overall Officials: Carly SY Lam, phD, Principal Investigator — School of Optometry, The Hong Kong Polytechnic University
Locations (1):
- The Centre of Myopia Ressearch, School of Optometry, The Hong Kong PolyU, Hong Kong, China